CLINICAL TRIAL: NCT06111092
Title: Testing Design Thinking Methodology to Engage Hispanic and Latino Families of Autistic Children in Research.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022C2-28939
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder; Patient Engagement
Keywords: Autism; Patient engagement
MeSH Terms: conditions — Autism Spectrum Disorder; Patient Participation; Autistic Disorder | interventions — Focus Groups

STUDY DESIGN:
Intervention Model Description: The aim of this study is to improve the health and well-being of Hispanic/Latino autistic children by improving the utilization of the evidence-based autism intervention Ayres Sensory Integration and to improve stakeholder engagement in the research process for effective outcomes. Specific aims of this project are:
  1. Compare DT and FG on measures of stakeholder engagement
  2. Compare the acceptability and feasibility of the adapted intervention manuals (one based on FG and another on DT data).
  Design: A randomized mixed methods design is used to evaluate stakeholder engagement. Phase one will compare two stakeholder engagement methods (Design Thinking -DT, and Focus Group - FG) and evaluate stakeholder engagement. Phase two uses data from phase one to culturally adapt the intervention (two separate intervention protocols will be adapted, one from FG data and another from DT data) and obtain stakeholder input on acceptability and feasibility for the Hispanic/Latino population
Who Masked: Participant, Outcomes Assessor
Masking Description: * data analysts are blind to the study arm so that their interpretation and analysis of the data is unbiased.
  * in Aim 2, the two adapted intervention protocols will be created, each based on data from either the design thinking or focus group sessions. These protocols will then be rated for acceptability, feasibility and cultural appropriateness using standardized measures and stakeholder input. This rating will be performed by individuals who are blinded to study arm that was used for adaptation of each protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Design Thinking Group (Other): A group of randomized participants (autistic adults, parents/caregivers, OT practitioners, teachers, and cultural experts) will participate in the Design Thinking (DT) process.
  Interventions: Other: Design Thinking
- Focus Group (Other): A group of randomized participants (autistic adults, parents/caregivers, OT practitioners, teachers, and cultural experts) will participate in the Focus Group (FG) process.
  Interventions: Other: Focus Groups

INTERVENTIONS:
Other: Design Thinking — Participants attend the DT session through all the stages that include emphasize, define, ideate, prototype and test.
  Arms: Design Thinking Group
Other: Focus Groups — Participants attend the FG that includes the introduction. discussion, and reflection.
  Arms: Focus Group

SUMMARY:
The goal of this study is to compare the level of engagement in the Hispanic and Latino parents of autistic children and culturally adapt the protocol of Ayres Sensory Integration to improve participation and health outcomes.

The main questions it aims to answer are:

Does the Design Thinking process result in higher stakeholder engagement and satisfaction in the research process in comparison to Focus Groups? Secondary question: Do cultural adaption using DT data yield higher scores of acceptability and implementation feasibility in comparison to FG methods?

Participants will:

* Be randomized into two groups of engagement (focus groups and design thinking)
* Be blinded (clinicians, selected caregivers, autistic persons, and cultural experts) and will rate the acceptability, feasibility, and cultural appropriateness of the protocol based on DT data higher than the protocol based on FG data.

DETAILED DESCRIPTION:
Racial and ethnic minorities with autistic children experience delays in access to therapy services that can result in poorer outcomes, decreased quality of life, and increased parental and financial stress. Many autism interventions were developed and tested with only White participants, assuming they could be transferable to minority populations. However, research has found that this is not the case and that interventions that are not adapted to an individual's culture and ethnicity do not work as well and are not used as frequently. In this project, we compare two methods of stakeholder engagement, Design Thinking (DT) and Focus Groups (FG), to determine which is better at getting input on the facilitators and barriers to access therapy for autistic children. We focus on Hispanics and Latinos as this is the largest minority group in the US, with one of the fastest-growing groups of autistic children. Our long-term objective is to improve the functional skills and health of Hispanic/Latino autistic children and their families by improving access to an occupational therapy intervention designed to improve daily living skills, socialization, and quality of life. Occupational therapy using Ayres Sensory Integration (OT/ASI) is the only evidence-based intervention that addresses the sensory symptoms in autism. We will use input from these engagement sessions to adapt two versions of the OT/ASI manual: one using DT data and the other using FG data. Outcomes are evaluated following each step. Following the completion of this project, the planned outputs of the study are data on the most effective minority stakeholder engagement method and a culturally adapted OT/ASI manual for Hispanic and Latino autistic children for clinicians and researchers. This information can support future researchers who are engaging Hispanic/Latino individuals or other minority groups in research.

Methods: A randomized mixed methods design is used to evaluate stakeholder engagement methods. Phase one will compare two stakeholder engagement methods (Design Thinking -DT, and Focus Group - FG) and evaluate stakeholder engagement based on the PCORI areas of stakeholder engagement which are operationalized in the Stakeholder-Centric Engagement Evaluation and qualitative data. Phase two utilizes data from phase one to culturally adapt the intervention (two separate intervention protocols will be adapted - one based on FG data and another based on DT data as described below), and obtain stakeholder input on acceptability and feasibility for the Hispanic/Latino autistic population. This provides a second way to measure the effectiveness of each stakeholder engagement method as we will have data to indicate which method (DT or FG) resulted in the highest-rated protocol. The data provided by this study will be used as a basis for a later comparative effectiveness study that will study the culturally adapted protocol's outcomes.

All sessions will be held in Spanish and/or English based on the groups' preferences. Since our intent is to hear the voices of Hispanic/Latino stakeholders, it seems valuable to hold focus groups in Spanish when the participants are Spanish as first language speakers (hereafter referred to as Spanish-first) with audio recordings and later transcription into English for analysis. To accommodate those who prefer English, we will make every effort to group these participants together. When, and if, the Spanish-first groups include participants who prefer English, we will have a Spanish to English translator available. In other words, we will be respectful of each participant's language to optimize their comfort in the engagement sessions.

This project addresses an urgent need to engage stakeholders as part of the research process from conceptualization to dissemination and the need for culturally sensitive evidence-based interventions for Hispanic/Latino autistic children. This project is being developed by a skilled and experienced team of investigators.

ELIGIBILITY:
Inclusion Criteria:

* Autistic person:

  * confirmed diagnosis of autism spectrum disorder
  * Hispanic/Latino
  * received therapeutic services as a child; and
  * willing and able (with i.e., language and cognitive skills) to participate in the design thinking or focus group session designed to learn about the facilitator and barriers to receipt of therapeutic services.
* Parent/caregiver:

  * Hispanic/Latino caregiver of an autistic child who receives or received therapeutic services such as occupational, physical, speech and language therapy
  * willing to participate in the design thinking or focus group session designed to learn about the facilitator and barriers to receipt of therapeutic services.
* Exclusion Criteria:

  * Do not meet age for autistic individual or diagnostic criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Stakeholder-Centric Engagement Evaluation | up to 14 weeks
  The instrument evaluates stakeholder engagement via the PCORI engagement principles. DT and FG participants use this instrument to rate engagement in throughout the research process using a Likert scale with 1= never and 5 = always.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM) and the Feasibility of Intervention Measure (FIM) (Weiner et al., 2017) | up to 14 weeks
  These are outcome measures that evaluate implementation success via the extent to which stakeholders believe the intervention is acceptable, appropriate, and feasible. Each measure uses a Likert response scale where 1 = completely disagree and 5 = completely agree.

CONTACTS AND LOCATIONS:
Overall Officials: Roseann C Schaaf, Principal Investigator — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: Yes
Publication in high-impact autism Journal and presentation at national and international autism research meetings.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following completion of the study and publication of findings.
Access Criteria: Upon written request (reviewed by the principal investigator) information will be shared.